CLINICAL TRIAL: NCT04663113
Title: Investigation of the Effect of Exercise Protocol Determined According to Metabolic Rate in Early Burn Patients on Coagulation, Fibrinolytic Activity and Functional Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Murat Ali ÇINAR, Resarch Asistant, Physical Therapist, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAC2020
Record Dates: First submitted 2020-11-16; First posted 2020-12-10 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Burns
Keywords: physiotherapy; Burn rehabilitation; Major burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: A total of 30 patients, 10 patients for each group, were planned to be included in the study.
  The individuals participating in the study will be divided into 3 groups: Standard therapy (1st Group), Standard therapy + bicycle ergometer (2nd Group) and Standard therapy + exercise protocol to be developed (3rd Group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): Standard physiotherapy (1st Group): It comprised of parameters such as early mobilization and ambulatory training, pulmonary physiotherapy, active and passive normal joint movement exercises.
  Interventions: Other: Control Group/1st group ( standard physiotherapy
- Aerobic Exercises group (Experimental): Aerobic exercise will be given with bicycle ergometer in addition to Standard physiotherapy (It comprised of parameters such as early mobilization and ambulatory training, pulmonary physiotherapy, active and passive normal joint movement exercises)
  Interventions: Other: 2nd group- Standard physiotherapy + bicycle ergometer
- the group in which the exercise protocol to be developed was applied (Experimental): Standard physiotherapy + exercise protocol to be developed: In addition to standard therapy, exercise will be given according to the measured basal metabolic rate of the patients.
  Interventions: Other: 3rd group- Standard physiotherapy + exercise protocol to be developed

INTERVENTIONS:
Other: Control Group/1st group ( standard physiotherapy — It comprised of parameters such as early mobilization and ambulatory training, pulmonary physiotherapy, active and passive normal joint movement exercises.
  Arms: Control group
Other: 2nd group- Standard physiotherapy + bicycle ergometer — Standard physiotherapy + bicycle ergometer: In addition to the standard therapy, a bicycle ergometer for 20 minutes 5 days a week will be given.
  Patients will turn the pedals of the bicycle while sitting on the edge of the bed.
  In this protocol, a portable bicycle with adjustable pedal system, which can be placed on the edge of the bed, will be used.
  "Ratings of perceived exertion (RPE)" will be used to determine the intensity of aerobic activity. According to the RPE, 10-12 strength exercises will be given.
  Arms: Aerobic Exercises group
Other: 3rd group- Standard physiotherapy + exercise protocol to be developed — Standard physiotherapy + exercise protocol to be developed: In addition to standard therapy, exercise will be given according to the measured basal metabolic rate of the patients.
  Portable indirect calorimetry will be used to measure the basal metabolic rates of the patients.
  The basal metabolic rates of the patients will be measured before the exercise and aerobic exercise or resistant exercise will be given according to the metabolic state of the patient.
  Ratings of perceived exertion (RPE) will be used as the aerobic exercise protocol and a 10-11 strength exercise will be given according to the RPE.
  If resistance exercise will be given, the intensity of the exercise (12-14) will be determined according to the RPE. Sandbags attached to the ankle will be used as a resistance exercise and 9 exercises were determined. (Knee extension, knee flexion, trunk flexion, trunk extension, hip extension, hip flexion, hip abduction, shoulder flexion, shoulder abduction
  Arms: the group in which the exercise protocol to be developed was applied

SUMMARY:
The aim of this study is; To investigate the Effect of the Exercise Protocol Determined According to Metabolic Rate in Early Burn Patients on Coagulation, Fibrinolytic Activity and Functional Capacity, and to create an exercise protocol that can guide researchers working in burn patients and physiotherapists working in burn centers at national and international level.

The study, which is planned to be carried out in Hasan Kalyoncu University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, will be included in the burn patients in the 25 Aralık State Hospital Burn Center, service and intensive care unit.

DETAILED DESCRIPTION:
Burn injury is one of the longest traumas, causing serious mortality and morbidity, and the length of hospital stay and rehabilitation period.

For optimal treatment after burns, all pathophysiological changes that may occur locally and systemically after injury should be well known.

Along with surgical and medical treatments, the role of early exercise in burn treatment is becoming more and more important.

Burn patients need a long rehabilitation period, including the acute period and the post-discharge period.

Early exercise is very important, especially in burn intensive care units, for healing of burns and minimizing the effects of hypermetabolism. Exercises should be started from the first day the patient is hospitalized.

In a study on physiotherapists working in 6 major burn centers in the United States, stated that all physiotherapists applied various exercises in the early period in burn patients, but these exercises varied in all centers in terms of characteristics such as type and frequency. In the same study, it was emphasized that exercise programs, which are the biggest help in reducing intensive care periods in burn patients, should be more consistent and there is a need for studies investigating the components of the exercises.

Stated in another study that the exercise program applied in the early period in burns does not have an internationally accepted standard and studies should be done to create an exercise prescription.

In recent years, it has been emphasized that exercise protocols differ between physiotherapists and that there is no international standardization in questionnaire studies on exercise protocols applied to burn patients.

In addition, it has been emphasized that studies investigating exercise components will contribute more to the burn literature.

The aim of this study is; To investigate the Effect of the Exercise Protocol Determined According to Metabolic Rate in Early Burn Patients on Coagulation, Fibrinolytic Activity and Functional Capacity, and to create an exercise protocol that can guide researchers working in burn patients and physiotherapists working in burn centers at national and international level.

The study, which is planned to be carried out in Hasan Kalyoncu University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, will be included in the burn patients in the 25 Aralık State Hospital Burn Center, service and intensive care unit.

Inclusion criteria

* Conscious patients
* Enterally fed
* >18 years old Exclusion criteria
* With inhalation burn
* In addition to existing burn trauma, those with other trauma (fracture, loss of limb, etc.)
* Organ dysfunctions or multiple organ failure
* History of chronic diseases such as diabetes, cholesterol and blood pressure
* prothrombin time> 14.6 sec A total of 30 patients, 10 patients for each group, were planned to be included in the study.

The individuals participating in the study will be divided into 3 groups: Standard therapy (1st Group), Standard therapy + bicycle ergometer (2nd Group) and Standard therapy + exercise protocol to be developed (3rd Group)

Assessment of Coagulation and Fibrinolytic Activity

Prothrombin time Platelet D-dimer, Fibrinogen

These parameters will be monitored 3 days a week for 6 weeks (These parameters will be monitored 3 days a week for 6 weeks (These biochemistry parameters are routinely checked in every patient at the 25 December State Hospital Burn Center)

Evaluation of Functional Capacity 6 min walking test Physiological consumption index MRC scale (general muscle strength measurement scale used in intensive care patients)

These parameters will be monitored weekly (once a week) for 6 weeks.

Evaluation of Basal Metabolism

For basal metabolism, "hand held device" indirect calorimeter will be used and individuals in each group will be evaluated and monitored daily.

ELIGIBILITY:
Inclusion Criteria:

Conscious patients Enterally fed >18 years old

Exclusion Criteria:

* With inhalation burn
* In addition to existing burn trauma, those with other trauma (fracture, loss of limb, etc.)
* Organ dysfunctions or multiple organ failure
* History of chronic diseases such as diabetes, cholesterol and blood pressure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
D-dimer (To measure coagulation changes and Fibrinolytic Activity) | Each participant will be evaluated for 6 weeks.
  blood test
fibrinogen (to measure changes in both coagulation and fibrinolytic activity) | Each participant will be evaluated for 6 weeks.
  blood test
prothrombin time | Each participant will be evaluated for 6 weeks.
  blood test
platelets (to measure changes in both coagulation and fibrinolytic activity) | Each participant will be evaluated for 6 weeks.
  blood test
6 min walking test | Each participant will be evaluated for 6 weeks.
  The test involves asking the patient to walk the longest distance possible in a set interval of 6 min, through a walking course (corridor) preferably 30-m long. healthy subjects, the 6-min walk distance(6MWD) ranges from 400 to 700 m
physiological consumption index | Each participant will be evaluated for 6 weeks.
  Physiological consumption index (PCI) was calculated ((walking heart rate) - (resting heart rate)) / (walking speed)]. 1
MRC scale ( Manaul muscle test) | Each participant will be evaluated for 6 weeks.
  Peripheral muscle strength of the upper and lower extremities will be measured manually with the Medical Research Council (MRC) scale and the Modified Medical Research Council 4-point scale (MMRC). Shoulder abduction, elbow flexion and wrist extension of the upper extremity; If it belongs to the lower extremity, hip flexion, knee extension and ankle dorsi flexion will be measured in the in-bed high sitting position as a modified position specific to intensive care. Grading according to the MRC scale is between 0-5 for each muscle group: the total MRC score is between 0-60, and values below 48 indicate muscle weakness.

CONTACTS AND LOCATIONS:
Overall Officials: Murat A ÇINAR, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veldema J, Bosl K, Kugler P, Ponfick M, Gdynia HJ, Nowak DA. Cycle ergometer training vs resistance training in ICU-acquired weakness. Acta Neurol Scand. 2019 Jul;140(1):62-71. doi: 10.1111/ane.13102. Epub 2019 May 10. PMID 30977897
- [Background] Keck M, Herndon DH, Kamolz LP, Frey M, Jeschke MG. Pathophysiology of burns. Wien Med Wochenschr. 2009;159(13-14):327-36. doi: 10.1007/s10354-009-0651-2. PMID 19652939
- [Background] Serghiou M, Cowan A, Whitehead C. Rehabilitation after a burn injury. Clin Plast Surg. 2009 Oct;36(4):675-86. doi: 10.1016/j.cps.2009.05.008. PMID 19793561
- [Result] Brusselaers N, Monstrey S, Vogelaers D, Hoste E, Blot S. Severe burn injury in Europe: a systematic review of the incidence, etiology, morbidity, and mortality. Crit Care. 2010;14(5):R188. doi: 10.1186/cc9300. Epub 2010 Oct 19. PMID 20958968
- [Result] Cinar MA, Bayramlar K, Erkilic A, Gunes A, Yakut Y. The effects of early physiotherapy on biochemical parameters in major burn patients: A burn center's experience. Ulus Travma Acil Cerrahi Derg. 2019 Sep;25(5):461-466. doi: 10.5505/tjtes.2018.05950. PMID 31475319
- [Result] Glas GJ, Levi M, Schultz MJ. Coagulopathy and its management in patients with severe burns. J Thromb Haemost. 2016 May;14(5):865-74. doi: 10.1111/jth.13283. Epub 2016 Mar 23. PMID 26854881
- [Result] Flores O, Tyack Z, Stockton K, Paratz JD. The use of exercise in burns rehabilitation: A worldwide survey of practice. Burns. 2020 Mar;46(2):322-332. doi: 10.1016/j.burns.2019.02.016. Epub 2019 Dec 18. PMID 31864784